CLINICAL TRIAL: NCT03793556
Title: Evaluation of the Effects of GERDOFF in Combination With a 6-week Therapy Based on Proton Pump Inhibitors Versus Proton Pump Inhibitors Alone on GERD-high Symptoms in Patients With Primary Diagnosis of Gastroesophageal Reflux Disease.
Brief Title: Evaluation of GERDOFF Efficacy in Combination With Proton Pump Inhibitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSC-DS GERD AP 16
Record Dates: First submitted 2018-12-11; First posted 2019-01-04 (Actual); Results first posted 2020-03-18 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Gastro-oesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole

STUDY DESIGN:
Intervention Model Description: Patients was randomized in an open-label treatment (in a ratio 1:1) and treated with the investigational medical device (IMD) + proton pump inhibitor (PPI) or PPI only for 6 weeks. At the end of treatment visit (V4) only patients who were classified as responders and belonging to the GERDOFF®+PPI group were included in the follow-up phase for 12 further weeks. During the follow-up, patients were randomized to an open-label treatment (in a 1:1 ratio) to GERDOFF® group or control group that will not receive any treatment for 12 weeks in order to evaluate the maintenance of treatment effects. To safeguard the health and well-being of patients, and to keep under control the possible upper symptoms of GERD that could appear, all patients that continued in the follow-up period received omeprazole as rescue medication, in a quantity adequate to cover the entire follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GERDOFF® + omeprazole (Experimental): GERDOFF® (tablets) was orally administered 3 times per day after meals; omeprazole was orally administered once a day before breakfast (2 capsules). The treatment lasted 6 weeks (+/- 2 days).
  Omeprazole was orally administered once a day before breakfast (2 capsules). The treatment lasted 6 weeks (+/- 2 days).
  Interventions: Device: GERDOFF® + Omeprazole
- Omeprazole (Active Comparator): Omeprazole was orally administered once a day before breakfast (2 capsules). The treatment lasted 6 weeks (+/- 2 days).
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Device: GERDOFF® + Omeprazole — GERDOFF® Hyaluronic acid + chondroitin sulphate + hydroxide aluminium Melt-in-mouth tablet 1100 mg + Omeprazole was orally administered once a day before breakfast (2 capsules). The treatment lasted 6 weeks (+/- 2 days).
  Other Names: GERDOFF®
  Arms: GERDOFF® + omeprazole
Drug: Omeprazole — Omeprazole, 2 capsules 20 mg, once a day before breakfast
  Other Names: Omeprazen
  Arms: Omeprazole

SUMMARY:
The aim of the present study was to evaluate the effect of a 6-weeks treatment of a CE-marked combination oral formulation of hyaluronic acid with chondroitin sulphate and aluminium hydroxide (GERDOFF®), in addition to proton pump inhibitors (PPI) at the standard dose, versus PPI only, in patients with first diagnosed clinical presentation of extra-esophageal GERD symptoms.

The investigators verified the reduction of symptoms frequency, using a Likert questionnaire, and severity, using the Reflux Symptom Index (RSI) questionnaire, to evaluate the proportion of Responders and Non-Responder patients in these two groups after 6 weeks of treatment, compared to baseline. Moreover investigators evaluated the persistence of effects of GERDOFF® + PPI treatment on extraesophageal symptoms, after a 12-weeks follow up, only in responder patients.

DETAILED DESCRIPTION:
Cough, hoarseness, prolonged voice lowering, and vocal timbre modification, without any documentable cause, are considered as minor disorders for which patients do not receive adequate attention. These disorders may represent extra-esophageal manifestations of gastro-oesophagea reflux. Accurate diagnosis and gastro-oesophageal reflux therapy have been proved as useful to improve patients' quality of life.

The aim of the present study was to evaluate, in first diagnosed patients presenting with upper symptoms associated with GERD, the effect of a 6-week treatment with a combination based on CS, HA and aluminium hydroxide (Gerdoff®), co-administered with a treatment with PPIs, compared to treatment with PPIs as monotherapy, i.e. to verify, in patients treated with the combination of the two products, the reduction in symptoms frequency by means of a Likert questionnaire and the severity of upper symptoms by means of the Reflux Symptom Index (RSI) questionnaire, and to collect safety data. After 6 weeks of treatment, patients included in the two groups were then classified as responders or non-responders. Responder patients were defined as those patients that, at the 6th week of treatment, reached a RSI score decreased for at least 50% compared to baseline and an absolute value < 13.

Furthermore, the maintenance of the effect of treatment on the extra-oesophageal symptoms was evaluated after a period of follow-up lasting 12 weeks, which could be entered only by responder patients randomised in the Gerdoff®-PPI arm. Patients included in the follow-up period were randomised to receive Gerdoff® or no treatment (control group). Safety data were also evaluated in the group of patients that continued in the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥ 18 years;
2. First diagnosis of GERD with upper symptoms, made on a clinical basis and confirmed by an ENT and/or confirmed by a Gastroenterologist using a RSI questionnaire;
3. Presence of extra-oesophageal symptoms associated with GERD;
4. RSI score ≥ 20;
5. Patients not pre-treated with PPIs, even for problems different from GERD, and/or with medical devices and/or similar products (e.g. antacid alginates etc..) in the last 4 weeks;
6. Cooperative patients, able to understand and adhere to the study procedures;
7. Patient able to freely give their written informed consent to study participation;
8. Patients that freely gave the consent to management of personal data related to the study.

Exclusion Criteria:

1. Known infective oesophagitis or oesophagitis due to acid or alkaline substances;
2. Acute or chronic rhinosinusitis;
3. Chronic bronchitis;
4. Known Zollinger-Ellison syndrome, hiatal hernia greater than 3 cm and Barrett oesophagus;
5. Ongoing neoplasias;
6. Uncontrolled diabetes;
7. Patients with impaired liver function;
8. Patients with rare hereditary problems of galactose intolerance;
9. Patients that, based on Investigator's opinion, could not take part in the study due to other diseases or concomitant therapies, such as the intake of atazanavir, nelfinavir, clopidogrel, posaconazole and erlotinib (as recommended in the Summary of Product Characteristics of Gerdoff®);
10. Patients with deficiency of Lapp lactase;
11. Patients with syndrome of glu-gal malabsorption;
12. Patients with hypersensitivity to omeprazole, substitute benzymidazolic or any of the excipients;
13. Patients already in treatment with PPIs or similar products;
14. Chronic use of drugs that interfere with the salivary secretion (e.g. anti-histamines or inhaled steroids);
15. Abuse of drug or alcohol;
16. Inability of the subject to adequately express his/her disturbances;
17. Patients with planned or ascertained pregnancy or that did not adopt an accepted contraceptive method;
18. Lactating patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- dr Alessandro Repici, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A first specialist visit was performed by an ENT as per clinical practice based on patient's symptoms.
  Patients sent by the ENT should not have been pre-treated with PPIs and/or medical devices and/or similar products. The diagnosis was confirmed by the Gastroenterologist Investigator who recruited patients.
Pre-assignment Details: In this phase of the study, 72 patients were enrolled. One patient withdrew the informed consent and was excluded from the study before randomization.
Groups:
- GERDOFF® + Omeprazole: GERDOFF® (tablets) was orally administered 3 times per day after meals; omeprazole was orally administered once a day before breakfast (2 capsules). The treatment lasted 6 weeks (+/- 2 days).
  GERDOFF®: GERDOFF® Hyaluronic acid + chondroitin sulphate + hydroxide aluminium Melt-in-mouth tablet 1100 mg
Period: Overall Study
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Started | 35 | 36
Completed | 22 | 34
Not Completed | 13 | 2
Not completed — Withdrawal by Subject | 12 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GERDOFF® + Omeprazole | Omeprazole | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Continuous [Median (Full Range); unit: years] | 46.0 [20 to 86] | 45.0 [20 to 76] | 46.0 [20 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 32 | 54
  Male | 13 | 4 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 36 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Patients with simultaneous symptoms [Number; unit: participants]
  1 symptom | 2 | 3 | 5
  2 symptoms | 5 | 1 | 6
  3 symptoms | 9 | 6 | 15
  4 symptoms | 11 | 17 | 28
  5 symptoms | 5 | 5 | 10
  6 symptoms | 2 | 3 | 5
  7 symptoms | 1 | 1 | 2
Hoarseness or vocal problem [Number; unit: participants]
  yes | 21 | 18 | 39
  no | 14 | 18 | 32
Throat clearance [Number; unit: participants]
  yes | 18 | 23 | 41
  no | 17 | 13 | 30
Excess of mucus in the throat or retrosternal fall of secretions [Number; unit: participants]
  yes | 14 | 15 | 29
  no | 21 | 21 | 42
Difficulty in swallowing food, fluids or pills [Number; unit: participants]
  yes | 7 | 7 | 14
  no | 28 | 29 | 57
Cough after the meal or after lying [Number; unit: participants]
  yes | 13 | 15 | 28
  no | 22 | 21 | 43
Difficulty in breathing or episodes of choking [Number; unit: participants]
  yes | 4 | 5 | 9
  no | 31 | 31 | 62
Problematic or troublesome cough [Number; unit: participants]
  yes | 16 | 12 | 28
  no | 19 | 24 | 43
Sensation of something blocked or mass in the throat [Number; unit: participants]
  yes | 17 | 12 | 29
  no | 18 | 24 | 42
Stomach burning, thoracic pain, poor digestion of gastric acid that moves upright [Number; unit: participants]
  yes | 17 | 22 | 39
  no | 18 | 14 | 32
Weight [Median (Full Range); unit: kg] — Population: Some data are missing in both arms
  kg
    number analyzed (Participants) | 29 | 31 | 60
    (all) | 63.0 [45.0 to 98.6] | 62.0 [43.0 to 95.0] | 62.5 [43 to 98.6]
Body Mass Index [Median (Full Range); unit: kg/m^2] — Population: Some data are missing in both arms
  kg/m^2
    number analyzed (Participants) | 29 | 31 | 60
    (all) | 22.6 [17.6 to 35.2] | 22.7 [16.8 to 38.6] | 22.7 [16.8 to 38.6]
Number of symptoms [Median (Full Range); unit: Symptom] | 4 [1 to 7] | 4 [1 to 7] | 4 [1 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Visit V4 of the Total Score of RSI Questionnaire
Description: After 6 weeks of treatment, the changes from baseline in the score of Reflux Symptom Index questionnaire were evaluated to verify the effects of treatments on high symptoms. The RSI questionnaire examines 9 items that are scored from 0 to 5, with a higher score that indicates a higher severity of the symptom (range of total score: 0-45).
Time Frame: In the first visit (baseline) and in the visit 4 (after 6 weeks of treatment)
Population: Four patients in the GERFOFF + omeprazole group did not complete the Reflux Symptom Index questionnaire and could not be included in the analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
Score on a scale | -16.2 (7.45) | -13.7 (10.58)
Statistical Analysis 1: Comparison: GERDOFF® + Omeprazole vs Omeprazole; Test type: Other; p = 0.276, Unpaired t test; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-7.03 to 2.04], Standard Deviation 9.27

2. Secondary Outcome: Total Score of Reflux Symptom Index Questionnaire in All Time-points Assessed
Description: Total score of the Reflux Symptom Index questionnaire assessed in all time-points.
  The RSI questionnaire examines 9 items, that are scored from 0 to 5, with a higher score that indicates a higher severity of the symptom (range of total score: 0-45).
Time Frame: In baseline Visit, Visit 2 (after 1 week), Visit 3 (after 3 weeks) and Visit 4 (after 6 weeks of treatment)
Population: Some data are missing; therefore, the number of participants in one or more rows differs from overall number analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 35 | 36
score on a scale
  Baseline | 24.2 (5.18) | 26.0 (4.96)
  Visit 2: number analyzed (Participants) | 32 | 35
  Visit 2 | 15.3 (7.86) | 19.6 (7.20)
  Visit 3: number analyzed (Participants) | 28 | 35
  Visit 3 | 12.9 (7.77) | 15.3 (8.08)
  Visit 4: number analyzed (Participants) | 31 | 36
  Visit 4 | 7.9 (6.04) | 12.3 (8.98)
Statistical Analysis 1: Comparison: GERDOFF® + Omeprazole vs Omeprazole; Test type: Other; p = 0.0157, ANOVA; The ANOVA model examined the entire curve profile

3. Secondary Outcome: Score of Hoarseness or Vocal Problem of the RSI Questionnaire Measured at the Baseline and in the Visit 4
Description: The Reflux Symptom Index questionnaire examines 9 items, including hoarseness or vocal problem that is score from 0 to 5, with a higher score that indicates a higher severity of the symptom.
Time Frame: At baseline and in the visit 4, after 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
score on a scale
  Baseline | 3.2 (1.35) | 2.8 (1.54)
  Visit 4 | 1.1 (1.33) | 1.6 (1.54)

4. Secondary Outcome: Score of Throat of the RSI Questionnarie Measured at the Baseline and in the Visit 4 of the RSI Questionnaire Score of Throat Clearance
Description: The Reflux Symptom Index questionnaire examines 9 items, including throat that is score from 0 to 5, with a higher score that indicates a higher severity of the symptom.
Time Frame: At baseline and in the visit 4, after 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
score on a scale
  Baseline | 3.4 (1.22) | 3.6 (1.00)
  Visit 4 | 1.4 (1.39) | 1.8 (1.37)

5. Secondary Outcome: Score of Excess of Mucus in the Throat or Retrosternal Fall of Secretions of the RSI Questionnaire Measured at Baseline and in the Visit 4
Description: The Reflux Symptom Index questionnaire examines 9 items, including excess of mucus in the throat or retrosternal fall of secretions that is score from 0 to 5, with a higher score that indicates a higher severity of the symptom.
Time Frame: At baseline and in the visit 4, after 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- GERDOFF® + Omeprazole: GERDOFF® (tablets) was orally administered 3 times per day after meals; omeprazole was orally administered once a day before breakfast (2 capsules). The treatment will last 6 weeks (+/- 2 days).
  GERDOFF®: GERDOFF® Hyaluronic acid + chondroitin sulphate + hydroxide aluminium Melt-in-mouth tablet 1100 mg
- Omeprazole: Omeprazole was orally administered once a day before breakfast (2 capsules). The treatment will last 6 weeks (+/- 2 days).
  Omeprazole: Omeprazole, 2 capsules 20 mg, once a day before breakfast
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
score on a scale
  Baseline | 2.7 (1.76) | 2.8 (1.77)
  Visit 4 | 1.4 (1.31) | 1.9 (1.61)

6. Secondary Outcome: Score of Difficulty in Swallowing Food, Fluids or Pills of the RSI Questionnaire Measured at Baseline and in the Visit 4
Description: The Reflux Symptom Index questionnaire examines 9 items, including difficulty in swallowing food, fluids or pills that is score from 0 to 5, with a higher score that indicates a higher severity of the symptom.
Time Frame: At baseline and in the visit 4, after 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
score on a scale
  Baseline | 1.9 (1.66) | 1.9 (1.84)
  Visit 4 | 0.4 (0.71) | 0.6 (0.94)

7. Secondary Outcome: Score of Cough of the RSI Questionnaire Measured at Baseline and in the Visit 4 After the Meal or After Lying
Description: The Reflux Symptom Index questionnaire examines 9 items, including cough that is score from 0 to 5, with a higher score that indicates a higher severity of the symptom.
Time Frame: At baseline and in the visit 4, after 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
score on a scale
  Baseline | 2.5 (1.76) | 3.3 (1.44)
  Visit 4 | 0.7 (1.01) | 1.7 (1.47)

8. Secondary Outcome: Score of Difficulty in Breathing or Episodes of Choking of the RSI Questionnaire Measured at Baseline and in the Visit 4
Description: The Reflux Symptom Index questionnaire examines 9 items, including difficulty in breathing or episodes of choking that is score from 0 to 5, with a higher score that indicates a higher severity of the symptom.
Time Frame: At baseline and in the visit 4, after 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
score on a scale
  Baseline | 1.5 (1.60) | 1.9 (1.69)
  Visit 4 | 0.5 (1.15) | 0.6 (0.97)

9. Secondary Outcome: Score of Problematic or Troublesome Cough of the RSI Questionnaire Measured at Baseline and in the Visit 4
Description: The Reflux Symptom Index questionnaire examines 9 items, including problematic or troublesome cough that is score from 0 to 5, with a higher score that indicates a higher severity of the symptom.
Time Frame: At baseline and in the visit 4, after 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
score on a scale
  Baseline | 2.5 (1.65) | 3.7 (1.19)
  Visit 4 | 0.8 (1.17) | 1.5 (1.54)

10. Secondary Outcome: Score of Sensation of Something Blocked or Mass in the Throat of the RSI Questionnaire Measured at Baseline and in the Visit 4
Description: The Reflux Symptom Index questionnaire examines 9 items, including sensation of something blocked or mass in the throat that is score from 0 to 5, with a higher score that indicates a higher severity of the symptom.
Time Frame: At baseline and in the visit 4, after 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
score on a scale
  Baseline | 3.0 (1.52) | 2.6 (1.75)
  Visit 4 | 0.8 (1.08) | 1.6 (1.59)

11. Secondary Outcome: Score of Stomach Burning, Thoracic Pain, Poor Digestion of Gastric Acid That Moves Upright of the RSI Questionnaire Measured at Baseline and in the Visit 4
Description: The Reflux Symptom Index questionnaire examines 9 items, including stomach burning, thoracic pain, poor digestion of gastric acid that moves upright that is score from 0 to 5, with a higher score that indicates a higher severity of the symptom.
Time Frame: At baseline and in the visit 4, after 6 weeks of treatment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
Score on a scale
  Baseline | 3.4 (1.56) | 3.5 (1.83)
  Visit 4 | 0.8 (1.08) | 3.5 (1.83)

12. Secondary Outcome: Number of Responders V4
Description: A responder was defined as a patient who at the 6th week of treatment showed a reduction of at least 50% vs. the baseline and an absolute value < 13 on the RSI questionnaire.
Time Frame: At visit 4 after 6 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
Participants
  Yes | 23 | 20
  No | 8 | 16
Statistical Analysis 1: Comparison: GERDOFF® + Omeprazole vs Omeprazole; Test type: Other; p = 0.0496, Chi-squared

13. Secondary Outcome: Number of Responders V6
Description: Responder patients of Group Gerdoff® + omeprazole were randomly assigned to receive a treatment with Gerdoff®-one tablet three times daily- All patients received a packaging of omeprazole, to be taken only if necessary, at constant dose and according to the indications of the Investigator. The scheduled duration of the follow-up period was 12 weeks.
  A responder was defined as a patient who at the 6th week of treatment showed a reduction of at least 50% vs. the baseline and an absolute value < 13 on the RSI questionnaire.
Time Frame: In the Visit 6 at the end of follow-up
Measure: Count of Participants; unit: Participants
Groups:
- No Treated: Responder patients of Group Gerdoff® + omeprazole were randomly assigned to the control group.
  All patients received a packaging of omeprazole, to be taken only if necessary, at constant dose and according to the indications of the Investigator. The scheduled duration of the follow-up period was 12 weeks.
Arm/Group | GERDOFF® + Omeprazole | No Treated
Number analyzed (Participants) | 9 | 8
Participants
  yes | 9 | 7
  No | 0 | 1

14. Secondary Outcome: Score of Upper Symptoms Using the Likert Scale at Baseline and in the Visit V4
Description: The Likert scale examines 9 symptoms, to be scored from 0 to 4, with a higher score indication a higher frequency of the symptom (i.e. 0=never, 1=occasionally, 2=sometimes, 3= often, 4=Always);
  The Likert scale scores of single items are as following:
  1. Hoarseness or vocal problem 0 1 2 3 4
  2. Throat clearance 0 1 2 3 4
  3. Excess of mucus in the throat or retrosternal fall of secretions 0 1 2 3 4
  4. Difficulty in swallowing food, fluids or pills 0 1 2 3 4
  5. Cough after the meal or after lying 0 1 2 3 4
  6. Difficulty in breathing or episodes of choking 0 1 2 3 4
  7. Problematic or troublesome cough 0 1 2 3 4
  8. Sensation of something blocked or mass in the throat 0 1 2 3 4
  9. Stomach burning, thoracic pain, poor digestion of gastric acid that moves upright 0 1 2 3 4.
  Subscales are summarized to compute a total score (total score ranges from 0-36). The mean values of Likert scale total score are reported.
Time Frame: At baseline and in the visit 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
Score on a scale
  Baseline | 19.0 (4.301) | 21 (4.557)
  Visit 4 | 7.4 (5.667) | 11.6 (8.083)
Statistical Analysis 1: Comparison: GERDOFF® + Omeprazole vs Omeprazole; Test type: Other; p = 0.0065, ANOVA

15. Secondary Outcome: Presence of Upper Symptoms at Visit 4, Using the RSI Questionnaire
Description: The Reflux Symptom Index questionnaire examines 9 items, to be scored from 0 to 5, with a higher score indication a higher severity of the symptom (range of total score: 0-45).
Time Frame: At visit 4 after weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
Participants
  Missing | 1 | 4
  1 symptom | 7 | 2
  2 symptoms | 6 | 9
  3 symptoms | 13 | 11
  4 symptoms | 4 | 7
  5 symptoms | 0 | 2
  6 symptoms | 0 | 1

16. Secondary Outcome: Use of Rescue Medication (Omeprazole) During the Treatment
Description: In the first 6 weeks of treatment, the intake in each treatment group of the rescue medication, allowed or not allowed, was calculated as the frequency of intake of the specific drug and the comparison between groups was performed using the Fisher's exact test.
Time Frame: From baseline to visit 4
Measure: Count of Participants; unit: Participants
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 35 | 36
Participants
  Yes | 24 | 28
  No | 11 | 8

17. Secondary Outcome: Use of Rescue Medication (Omeprazole) During the Follow-up
Description: During the follow-up, the intake in each treatment group of the rescue medication, allowed or not allowed, was calculated as the frequency of intake of the specific drug.
Time Frame: In the Visit 6 after 12 weeks from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | GERDOFF® + Omeprazole | No Treated
Number analyzed (Participants) | 9 | 8
Participants
  Yes | 7 | 5
  No | 2 | 3

18. Secondary Outcome: Use of Rescue Medication (Other Than Omeprazole) During Treatment
Description: During treatment, the intake in each treatment group of the rescue medication, allowed or not allowed, was calculated as the frequency of intake of the specific drug.
Time Frame: From baseline to visit 4
Measure: Count of Participants; unit: Participants
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
Participants
  Yes | 0 | 4
  No | 31 | 32

19. Secondary Outcome: Patients'Satisfaction
Description: This evaluation was expressed with a semi-quantitative ordinal scale: 0 = low, 1 = discrete, 2 = good, 3 = excellent).
Time Frame: At visit 4 after weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
Number analyzed (Participants) | 31 | 36
Participants
  Missing | 1 | 0
  Low | 3 | 1
  Discrete | 1 | 7
  Good | 11 | 11
  Excellent | 15 | 17

ADVERSE EVENTS:
Time Frame: During the 6 weeks of treatment in non-responders in the group GERDOFF+PPI and in patients randomized in PPI group; during the 6 weeks of treatment and 12-week follow-up in responder patients randomized in the group GERDOFF + PPI
Arm/Group | GERDOFF® + Omeprazole | Omeprazole
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/36
Other Adverse Events (participants affected / at risk) | 14/35 | 12/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GERDOFF® + Omeprazole (N=35) | Omeprazole (N=36)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GERDOFF® + Omeprazole (N=35) | Omeprazole (N=36)
Migraine (Nervous system disorders) | 2 (3) | 0 (0)
Flu-like symptoms (General disorders) | 3 (5) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Red blood cell sedimentation rate increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased subjects affected / exposed (Investigations) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Clonus (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysentery (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT03793556/Prot_SAP_000.pdf